CLINICAL TRIAL: NCT02843906
Title: Cognitive, Morphological and Neurobiological Progressive Aspects in Bipolar Disorders in the Elderly: Toward to a Neurodegenerescence Detection?
Acronym: BIPAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Tours (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Marseille (Other); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire de Besancon (Other); Central Hospital, Nancy, France (Other); University Hospital, Clermont-Ferrand (Other); Versailles Hospital (Other); University Hospital, Montpellier (Other); Reims University hospital (Other); Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 38RC13.217
Record Dates: First submitted 2016-05-11; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Senile Plaques; Tau Proteins; Alzheimer Disease; Bipolar Disorders; Mild Cognitive Impairment
Keywords: alzheimer disease; bipolar disorders; mild cognitive impairement
MeSH Terms: conditions — Plaque, Amyloid; Alzheimer Disease; Bipolar Disorder; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy; tetraethylpyrazine; Fluorodeoxyglucose F18; Neuropsychological Tests; Apolipoproteins; Apolipoproteins E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BD/CD + (Active Comparator): Lombar punction, RMI, TEP/FDG, ApoE detection, psychiatric tests, neuropsychological tests
  Interventions: Procedure: Lombar Punction; Radiation: Magnetic Resonance Imaging (MRI); Radiation: Positron-Emission Tomography (TEP) /(FDG); Other: Psychiatric tests; Other: Neuropsychological Tests; Genetic: Apolipoprotein (ApoE) detection
- BD/CD - (Active Comparator): Lombar punction, RMI, TEP/FDG, ApoE detection, psychiatric tests, neuropsychological tests
  Interventions: Procedure: Lombar Punction; Radiation: Magnetic Resonance Imaging (MRI); Radiation: Positron-Emission Tomography (TEP) /(FDG); Other: Psychiatric tests; Other: Neuropsychological Tests; Genetic: Apolipoprotein (ApoE) detection
- a-MCI (Active Comparator): Lombar punction, RMI, TEP/FDG, ApoE detection, psychiatric tests, neuropsychological tests
  Interventions: Procedure: Lombar Punction; Radiation: Magnetic Resonance Imaging (MRI); Radiation: Positron-Emission Tomography (TEP) /(FDG); Other: Psychiatric tests; Other: Neuropsychological Tests; Genetic: Apolipoprotein (ApoE) detection

INTERVENTIONS:
Procedure: Lombar Punction — cerebrospinal fluid testing at screening and M36
Radiation: Magnetic Resonance Imaging (MRI) — MRI done at screening and M36
Radiation: Positron-Emission Tomography (TEP) /(FDG) — TEP/FDG done at screening and M36
Other: Psychiatric tests
Other: Neuropsychological Tests — done at screening, M12, M24 and M36
Genetic: Apolipoprotein (ApoE) detection — ApoE detection done at screening

SUMMARY:
The purpose of this study is to identify association between cerebrospinal fluid Alzheimer's Disease's neurodegenerescence biomarkers (tau, ptau, Aß40 and Aß1-42) and occurrence of cognitive deficits in older patients with bipolar disorders.

ELIGIBILITY:
Inclusion Criteria:

* male or female subject aged between 60 and 80 years old
* in patient or out-patient at one of the centers participating in the study
* Mini-mental state examination (MMSE) score > 20 at baseline
* patient with diagnostic of amnestic-Mild Cognitive Impairment
* patients suffering of bipolar disorders type I or II
* in remitted (euthymic) state at baseline

Exclusion Criteria:

* pre-existing history of dementia
* history of neurologic disorder
* lifetime history of a severe psychiatric disorder other than bipolar disorders
* current medical problems
* patients treated with electroconvulsive therapy within the past six months
* patients with substance abuse or dependence within the past 12 months
* patients hospitalized without consent

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Functionnal/Cognitive evaluation | Half an hour
  Global cognitive evaluation :
  MMSE (Mini-Mental State Examination), CDR, BREF, 5 word of Dubois ADL, IADL.
Psychatric evaluation | 15 minutes
  Semi-directive psychiatric interview.
Psychatric evaluation | 15 minutes
  Scales for thymus evaluation : GDS, YMRS, BPRS, STAI
Brain MRI | 40 minutes
  Enable neuropsychological evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: BOUGEROL BT Thierry, Professor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Tours, Tours, France

REFERENCES:
- [Background] Ali SO, Denicoff KD, Altshuler LL, Hauser P, Li X, Conrad AJ, Smith-Jackson EE, Leverich GS, Post RM. Relationship between prior course of illness and neuroanatomic structures in bipolar disorder: a preliminary study. Neuropsychiatry Neuropsychol Behav Neurol. 2001 Oct-Dec;14(4):227-32. PMID 11725216
- [Background] Amieva H, Le Goff M, Millet X, Orgogozo JM, Peres K, Barberger-Gateau P, Jacqmin-Gadda H, Dartigues JF. Prodromal Alzheimer's disease: successive emergence of the clinical symptoms. Ann Neurol. 2008 Nov;64(5):492-8. doi: 10.1002/ana.21509. PMID 19067364
- [Background] Bora E, Vahip S, Gonul AS, Akdeniz F, Alkan M, Ogut M, Eryavuz A. Evidence for theory of mind deficits in euthymic patients with bipolar disorder. Acta Psychiatr Scand. 2005 Aug;112(2):110-6. doi: 10.1111/j.1600-0447.2005.00570.x. PMID 15992392
- [Background] Chetelat G, Eustache F, Viader F, De La Sayette V, Pelerin A, Mezenge F, Hannequin D, Dupuy B, Baron JC, Desgranges B. FDG-PET measurement is more accurate than neuropsychological assessments to predict global cognitive deterioration in patients with mild cognitive impairment. Neurocase. 2005 Feb;11(1):14-25. doi: 10.1080/13554790490896938. PMID 15804920
- [Background] Chetelat G, Desgranges B, Eustache F. [Brain profile of hypometabolism in early Alzheimer's disease: relationships with cognitive deficits and atrophy]. Rev Neurol (Paris). 2006 Oct;162(10):945-51. doi: 10.1016/s0035-3787(06)75104-9. French. PMID 17028562
- [Background] Corder EH, Saunders AM, Strittmatter WJ, Schmechel DE, Gaskell PC, Small GW, Roses AD, Haines JL, Pericak-Vance MA. Gene dose of apolipoprotein E type 4 allele and the risk of Alzheimer's disease in late onset families. Science. 1993 Aug 13;261(5123):921-3. doi: 10.1126/science.8346443.
- [Background] Delaloye C, Moy G, Baudois S, de Bilbao F, Remund CD, Hofer F, Ragno Paquier C, Campos L, Weber K, Gold G, Moussa A, Meiler CC, Giannakopoulos P. Cognitive features in euthymic bipolar patients in old age. Bipolar Disord. 2009 Nov;11(7):735-43. doi: 10.1111/j.1399-5618.2009.00741.x. Epub 2009 Aug 28. PMID 19719786
- [Background] Delaloye C, Moy G, de Bilbao F, Weber K, Baudois S, Haller S, Xekardaki A, Canuto A, Giardini U, Lovblad KO, Gold G, Giannakopoulos P. Longitudinal analysis of cognitive performances and structural brain changes in late-life bipolar disorder. Int J Geriatr Psychiatry. 2011 Dec;26(12):1309-18. doi: 10.1002/gps.2683. Epub 2011 Mar 10. PMID 21394788
- [Background] Doring TM, Kubo TT, Cruz LC Jr, Juruena MF, Fainberg J, Domingues RC, Gasparetto EL. Evaluation of hippocampal volume based on MR imaging in patients with bipolar affective disorder applying manual and automatic segmentation techniques. J Magn Reson Imaging. 2011 Mar;33(3):565-72. doi: 10.1002/jmri.22473. PMID 21563239
- [Background] Ewers M, Buerger K, Teipel SJ, Scheltens P, Schroder J, Zinkowski RP, Bouwman FH, Schonknecht P, Schoonenboom NS, Andreasen N, Wallin A, DeBernardis JF, Kerkman DJ, Heindl B, Blennow K, Hampel H. Multicenter assessment of CSF-phosphorylated tau for the prediction of conversion of MCI. Neurology. 2007 Dec 11;69(24):2205-12. doi: 10.1212/01.wnl.0000286944.22262.ff. PMID 18071141
- [Background] Fagan AM, Mintun MA, Shah AR, Aldea P, Roe CM, Mach RH, Marcus D, Morris JC, Holtzman DM. Cerebrospinal fluid tau and ptau(181) increase with cortical amyloid deposition in cognitively normal individuals: implications for future clinical trials of Alzheimer's disease. EMBO Mol Med. 2009 Nov;1(8-9):371-80. doi: 10.1002/emmm.200900048. PMID 20049742
- [Background] Hindley NJ, Jobst KA, King E, Barnetson L, Smith A, Haigh AM. High acceptability and low morbidity of diagnostic lumbar puncture in elderly subjects of mixed cognitive status. Acta Neurol Scand. 1995 May;91(5):405-11. doi: 10.1111/j.1600-0404.1995.tb07029.x. PMID 7639073
- [Background] Jones LD, Payne ME, Messer DF, Beyer JL, MacFall JR, Krishnan KR, Taylor WD. Temporal lobe volume in bipolar disorder: relationship with diagnosis and antipsychotic medication use. J Affect Disord. 2009 Apr;114(1-3):50-7. doi: 10.1016/j.jad.2008.07.003. Epub 2008 Aug 8. PMID 18691766
- [Background] Kessing LV, Nilsson FM. Increased risk of developing dementia in patients with major affective disorders compared to patients with other medical illnesses. J Affect Disord. 2003 Feb;73(3):261-9. doi: 10.1016/s0165-0327(02)00004-6. PMID 12547295
- [Background] Kessing LV, Andersen PK. Does the risk of developing dementia increase with the number of episodes in patients with depressive disorder and in patients with bipolar disorder? J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1662-6. doi: 10.1136/jnnp.2003.031773. PMID 15548477
- [Background] Li G, Sokal I, Quinn JF, Leverenz JB, Brodey M, Schellenberg GD, Kaye JA, Raskind MA, Zhang J, Peskind ER, Montine TJ. CSF tau/Abeta42 ratio for increased risk of mild cognitive impairment: a follow-up study. Neurology. 2007 Aug 14;69(7):631-9. doi: 10.1212/01.wnl.0000267428.62582.aa. PMID 17698783
- [Background] Masouy A, Chopard G, Vandel P, Magnin E, Rumbach L, Sechter D, Haffen E. Bipolar disorder and dementia: where is the link? Psychogeriatrics. 2011 Mar;11(1):60-7. doi: 10.1111/j.1479-8301.2010.00348.x. PMID 21447111
- [Background] Martino DJ, Igoa A, Marengo E, Scapola M, Ais ED, Strejilevich SA. Cognitive and motor features in elderly people with bipolar disorder. J Affect Disord. 2008 Jan;105(1-3):291-5. doi: 10.1016/j.jad.2007.05.014. Epub 2007 Jun 18. PMID 17573121
- [Background] Meeks S. Bipolar disorder in the latter half of life: symptom presentation, global functioning and age of onset. J Affect Disord. 1999 Jan-Mar;52(1-3):161-7. doi: 10.1016/s0165-0327(98)00069-x. PMID 10357029
- [Background] Peskind E, Nordberg A, Darreh-Shori T, Soininen H. Safety of lumbar puncture procedures in patients with Alzheimer's disease. Curr Alzheimer Res. 2009 Jun;6(3):290-2. doi: 10.2174/156720509788486509. PMID 19519311
- [Background] Peskind ER, Riekse R, Quinn JF, Kaye J, Clark CM, Farlow MR, Decarli C, Chabal C, Vavrek D, Raskind MA, Galasko D. Safety and acceptability of the research lumbar puncture. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19(4):220-5. doi: 10.1097/01.wad.0000194014.43575.fd. PMID 16327349
- [Background] Preuss UW, Watzke S, Choi JH. Diagnostic correlates of Alzheimer dementia in a U.S. Nationwide inpatient sample. Am J Geriatr Psychiatry. 2010 Sep;18(9):821-9. doi: 10.1097/JGP.0b013e3181ca3a13. PMID 20220586
- [Background] Saunders AM, Strittmatter WJ, Schmechel D, George-Hyslop PH, Pericak-Vance MA, Joo SH, Rosi BL, Gusella JF, Crapper-MacLachlan DR, Alberts MJ, et al. Association of apolipoprotein E allele epsilon 4 with late-onset familial and sporadic Alzheimer's disease. Neurology. 1993 Aug;43(8):1467-72. doi: 10.1212/wnl.43.8.1467. PMID 8350998
- [Background] Tapiola T, Alafuzoff I, Herukka SK, Parkkinen L, Hartikainen P, Soininen H, Pirttila T. Cerebrospinal fluid beta-amyloid 42 and tau proteins as biomarkers of Alzheimer-type pathologic changes in the brain. Arch Neurol. 2009 Mar;66(3):382-9. doi: 10.1001/archneurol.2008.596. PMID 19273758
- [Background] Thomann PA, Kaiser E, Schonknecht P, Pantel J, Essig M, Schroder J. Association of total tau and phosphorylated tau 181 protein levels in cerebrospinal fluid with cerebral atrophy in mild cognitive impairment and Alzheimer disease. J Psychiatry Neurosci. 2009 Mar;34(2):136-42. PMID 19270764
- [Background] Vemuri P, Wiste HJ, Weigand SD, Knopman DS, Trojanowski JQ, Shaw LM, Bernstein MA, Aisen PS, Weiner M, Petersen RC, Jack CR Jr; Alzheimer's Disease Neuroimaging Initiative. Serial MRI and CSF biomarkers in normal aging, MCI, and AD. Neurology. 2010 Jul 13;75(2):143-51. doi: 10.1212/WNL.0b013e3181e7ca82. PMID 20625167
- [Background] Verghese PB, Castellano JM, Holtzman DM. Apolipoprotein E in Alzheimer's disease and other neurological disorders. Lancet Neurol. 2011 Mar;10(3):241-52. doi: 10.1016/S1474-4422(10)70325-2. PMID 21349439
- [Background] Wingo AP, Harvey PD, Baldessarini RJ. Neurocognitive impairment in bipolar disorder patients: functional implications. Bipolar Disord. 2009 Mar;11(2):113-25. doi: 10.1111/j.1399-5618.2009.00665.x. PMID 19267694
- [Background] Zetterberg H, Tullhog K, Hansson O, Minthon L, Londos E, Blennow K. Low incidence of post-lumbar puncture headache in 1,089 consecutive memory clinic patients. Eur Neurol. 2010;63(6):326-30. doi: 10.1159/000311703. Epub 2010 Jun 3. PMID 20516693